CLINICAL TRIAL: NCT01216631
Title: Intra-articular and Intravenous Infliximab in the Treatment of Resistant Seronegative Oligoarthritis of the Knee
Brief Title: Seronegative Oligoarthritis of the Knee Study (SOKS)
Acronym: SOKS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to recruit
Sponsor: University of Leeds (Other)
Collaborators: Centocor, Inc. (Industry)
Responsible Party: Principal Investigator, Laura Coates, NIHR Clinical Lecturer, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-015810-23
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Results first posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Spondylarthropathies
Keywords: seronegative; oligoarthritis; infliximab; intraarticular
MeSH Terms: conditions — Spondylarthropathies; Arthritis | interventions — Methylprednisolone; Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- IA steroid (Active Comparator): Intra-articular injection of steroid (80mg depomedrone)
  Interventions: Drug: methylprednisolone
- IA infliximab (Experimental): intra-articular injection of 100mg infliximab
  Interventions: Drug: Infliximab
- IV infliximab (Experimental): intravenous infusions of infliximab given at 0, 2, 6 and 14 weeks at a dose of 5mg/kg (patient body weight)
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: methylprednisolone — intra-articular injection of methylprednisolone (80mg given at baseline only)
  Other Names: depomedrone
  Arms: IA steroid
Drug: Infliximab — intra-articular injection of 100mg infliximab given at baseline only
  Other Names: remicade
  Arms: IA infliximab
Drug: Infliximab — intravenous infliximab at a dose of 5mg/kg (as per patient weight) given at week 0, 2, 6 and 14
  Other Names: remicade
  Arms: IV infliximab

SUMMARY:
The aim of this study is to establish the efficacy and duration of effect of intra-articular (IA) infliximab vs intravenous infliximab vs current standard care (IA steroid injections) in seronegative oligoarthritis. All patients will have seronegative arthritis affecting less than 5 joints but including at least one knee. 10 patients will receive IA infliximab injections to the affected knee, 10 will receive IA steroid injections to the affected knee and 10 will receive a course of intravenous infliximab. Patients will not be aware of their group as this is a placebo-controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Inflammatory oligoarthritis (4 or less active joints) with at least one swollen knee joint of at least 3 months duration
* Rheumatoid factor and anti-CCP Ab negative
* Either arthritis onset at <45 years of age, or arthritis onset at ≥45 years of age with early morning stiffness>30mins or raised inflammatory markers
* If under 40 years of age, clinical exclusion of a diagnosis of gout.
* If 40 years or older at screening, a prior normal examination of synovial fluid from the affected joint excluding crystal arthropathy or infection.
* Failure of methotrexate (inefficacy after >3 month trial, intolerance or contra-indication)
* Have the capacity to understand and sign an informed consent form.
* Gender: male or female
* 18 years of age or over.
* Women must be either postmenopausal (no menstrual period for a minimum of 1 year) or surgically sterilized or in use of adequate birth control measures and have a negative serum pregnancy test on entry in the study.
* Men and women of childbearing potential must use adequate birth control measures (e.g., abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, implantable or injectable contraceptives or surgical sterilization) for the duration of the study and should continue such precautions for 6 months after receiving the last infusion.
* Are considered eligible according to the tuberculosis (TB) eligibility assessment, screening, and early detection of reactivation rules defined in the protocol
* The screening laboratory test results must meet the following criteria

  * WBC (white blood cell count): >3.5 x 109/L
  * ANC (absolute neutrophil count): >1.5 x 109/L
  * Hemoglobin: >10g/dL
  * Platelets: >120 x 109/L
  * SGPT (ALT - alanine aminotransferase) < 1.5 times upper normal limit (i.e. 60iu/L)
* Have no history of latent or active TB prior to screening. An exception is made for subjects with a history of latent TB and documentation of having completed appropriate treatment for latent TB (see Appendix 3) within 3 years prior to the first administration of study agent. It is the responsibility of the investigator to verify the adequacy of previous anti-tuberculous treatment and provide appropriate documentation.
* Have no signs or symptoms suggestive of active TB upon medical history and/or physical examination.
* Have had no recent close contact with a person with active TB or, if there has been such contact, will be referred to a physician specializing in TB to undergo additional evaluation and, if warranted, receive appropriate treatment for latent TB prior to the first administration of study agent.
* Within 6 weeks prior to the first administration of study agent, either have a negative QuantiFeron test result (see Appendix 3) or have a newly identified positive QuantiFeron test result during screening in which active TB has been ruled out and for which appropriate treatment for latent TB has been initiated prior to the first administration of study agent.
* Have a chest radiograph (posterior-anterior view and if required, a lateral view), taken within 3 months prior to the first administration of study agent and read by a qualified radiologist, with no evidence of current, active TB or old, inactive TB.

Exclusion Criteria:

* Grade 4 osteoarthritis (Kellgren-Lawrence score) on plain radiograph of the knee
* Rheumatoid Arthritis (defined by the ACR criteria for the diagnosis of RA, 1987)
* Ankylosing Spondylitis (defined by the modified New York Criteria)
* Clinical diagnosis of gout or previous evidence of crystal arthropathy on synovial fluid aspirates
* Women who are pregnant, nursing, or planning pregnancy within 6 months after the last infusion (this includes father's who plan on fathering a child within 6 months after their last infusion).
* Have had any previous treatment with biological therapies.
* History of receiving human/murine recombinant products or a known allergy to murine products. A known allergy to murine product is definitely an exclusion criterion
* Previous intra-muscular, intra-articular or intra-venous steroids within 4 weeks prior to baseline.
* Previous oral steroids at a dose >10mg/day prednisolone or equivalent for 4 weeks prior to baseline.
* Documentation of seropositive for human immunodeficiency virus (HIV).
* Documentation of a positive test for hepatitis B surface antigen or hepatitis C.
* Have a history of alcohol or substance abuse within the preceding 6 months that, in the opinion of the investigator, may increase the risks associated with study participation or study agent administration, or may interfere with interpretation of results.
* Have a known history of serious infections (e.g., hepatitis, pneumonia, or pyelonephritis) in the previous 3 months.
* Have or have had an opportunistic infection (e.g., herpes zoster [shingles], cytomegalovirus, Pneumocystis carinii, aspergillosis, histoplasmosis, or mycobacteria other than TB) within 6 months prior to screening
* Have had a Bacille Calmette-Guérin (BCG) vaccination within 12 months of screening.
* Are considered ineligible according to the TB eligibility assessment, screening, and early detection of reactivation rules described in Appendix 3.
* Have a chest radiograph within 3 months prior to the first administration of study agent that shows an abnormality suggestive of a malignancy or current active infection.
* Have a history of lymphoproliferative disease, including lymphoma or signs suggestive of possible lymphoproliferative disease such as lymphadenopathy of unusual size or location (e.g., nodes in the posterior triangle of the neck, infraclavicular, epitrochlear, or periaortic area), or splenomegaly.
* Currently have any known malignancy other than the condition being treated or have a history of malignancy, with the exception of basal cell or squamous cell carcinoma of the skin that has been fully excised with no evidence of recurrence.
* Have current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or cerebral disease.
* Are unable or unwilling to undergo multiple venipunctures because of poor tolerability or lack of easy access.
* Use of any investigational drug within 30 days prior to screening or within 5 half-lives of the investigational agent, whichever is longer.
* Presence of a transplanted solid organ (with the exception of a corneal transplant > 3 months prior to screening).
* Have a concomitant diagnosis or history of congestive heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip G Conaghan, FRCP, Principal Investigator — University of Leeds
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IA Steroid | IA Infliximab | IV Infliximab
Started | 0 | 0 | 1
Completed | 0 | 0 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only 1 recruited
Groups:
- Total: Total of all reporting groups
Arm/Group | IA Steroid | IA Infliximab | IV Infliximab | Total
Number analyzed (Participants) | 0 | 0 | 1 | 1
Age, Categorical [Number; unit: participants]
  <=18 years |  |  | 0 | 0
  Between 18 and 65 years |  |  | 1 | 1
  >=65 years |  |  | 0 | 0
Gender [Number; unit: participants]
  Female |  |  | 0 | 0
  Male |  |  | 1 | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom |  |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Ultrasound Synovitis Score
Description: reduction of ultrasound synovitis score of the affected knee at 8 weeks following intiation of treatment
Time Frame: 8 weeks
Population: Only one patient was recruited for this study due to problems with recruitment. Therefore outcome measure data is not analysed as only one patient was recruited.
Arm/Group | IA Steroid | IA Infliximab | IV Infliximab
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: US Synovitis Score
Description: Change in US synovitis score of the affected knee at 2 and 8 weeks after treatment initiation
Time Frame: 2 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Pain Visual Analogue Scale
Description: Change in patient's assessment of pain by a 100mm visual analogue score
Time Frame: 2 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Psoriatic Arthritis Quality of Life Scale (PsQOL)
Description: Change in PsQOL score from baseline
Time Frame: 2 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Rheumatoid Arthritis Outcome Score (RAOS)
Description: Change in RAOS questionnaire score
Time Frame: 2 weeks
Reporting Status: Not Posted

6. Secondary Outcome: US Synovitis Score
Description: Change in US synovitis score of the affected knee at 2 and 8 weeks after treatment initiation
Time Frame: 16 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Pain Visual Analogue Scale
Description: Change in patient's assessment of pain by a 100mm visual analogue score
Time Frame: 6 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Pain Visual Analogue Scale
Description: Change in patient's assessment of pain by a 100mm visual analogue score
Time Frame: 8 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Pain Visual Analogue Scale
Description: Change in patient's assessment of pain by a 100mm visual analogue score
Time Frame: 14 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Pain Visual Analogue Scale
Description: Change in patient's assessment of pain by a 100mm visual analogue score
Time Frame: 16 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Psoriatic Arthritis Quality of Life Scale (PsQOL)
Description: Change in PsQOL score from baseline
Time Frame: 26 weeks
Reporting Status: Not Posted

12. Secondary Outcome: Psoriatic Arthritis Quality of Life Scale (PsQOL)
Description: Change in PsQOL score from baseline
Time Frame: 6 weeks
Reporting Status: Not Posted

13. Secondary Outcome: Psoriatic Arthritis Quality of Life Scale (PsQOL)
Description: Change in PsQOL score from baseline
Time Frame: 8 weeks
Reporting Status: Not Posted

14. Secondary Outcome: Psoriatic Arthritis Quality of Life Scale (PsQOL)
Description: Change in PsQOL score from baseline
Time Frame: 14 weeks
Reporting Status: Not Posted

15. Secondary Outcome: Psoriatic Arthritis Quality of Life Scale (PsQOL)
Description: Change in PsQOL score from baseline
Time Frame: 16 weeks
Reporting Status: Not Posted

16. Secondary Outcome: Psoriatic Arthritis Quality of Life Scale (PsQOL)
Description: Change in PsQOL score from baseline
Time Frame: 26 weeks
Reporting Status: Not Posted

17. Secondary Outcome: Rheumatoid Arthritis Outcome Score (RAOS)
Description: Change in RAOS questionnaire score
Time Frame: 6 weeks
Reporting Status: Not Posted

18. Secondary Outcome: Rheumatoid Arthritis Outcome Score (RAOS)
Description: Change in RAOS questionnaire score
Time Frame: 8 weeks
Reporting Status: Not Posted

19. Secondary Outcome: Rheumatoid Arthritis Outcome Score (RAOS)
Description: Change in RAOS questionnaire score
Time Frame: 14 weeks
Reporting Status: Not Posted

20. Secondary Outcome: Rheumatoid Arthritis Outcome Score (RAOS)
Description: Change in RAOS questionnaire score
Time Frame: 16 weeks
Reporting Status: Not Posted

21. Secondary Outcome: Rheumatoid Arthritis Outcome Score (RAOS)
Description: Change in RAOS questionnaire score
Time Frame: 26 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | IA Steroid | IA Infliximab | IV Infliximab
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes